CLINICAL TRIAL: NCT05595343
Title: Learning Curves in Laparoscopic Distal Pancreatectomy: A Different Experience for Each Generation
Status: Completed | Type: Observational
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Other Study IDs: W19_414 # 19.482
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early adopting surgeons: Surgeons who started performing LDP during phase 3 of the IDEAL framework; the Assessment phase. They received training in the form of fellowships, proctoring, and courses
  Interventions: Procedure: Laparoscopic distal pancreatectomy
- Pioneering surgeons: Surgeons who started performing LDP during phase 2 of the IDEAL framework; the Development and Exploration phase. They did not receive any specific form of training and were therefore considered self-taught.
  Interventions: Procedure: Laparoscopic distal pancreatectomy

INTERVENTIONS:
Procedure: Laparoscopic distal pancreatectomy — Comparison of performed laparoscopic distal pancreas surgery in two different surgeon groups

SUMMARY:
This study compared the learning curves and outcome of Laparoscopic Distal Pancreatectomy between 'pioneers' and early adopters in terms of feasibility and proficiency using short term outcomes.

DETAILED DESCRIPTION:
Learning curves of laparoscopic distal pancreatectomy (LDP) are mostly based on 'pioneering' surgeons who acquired sufficient proficiency largely through self-teaching. No learning curves have been investigated for early adopting surgeons who performed surgery in later stages of the IDEAL framework and build on the experience of the 'pioneering' surgeons. This study compared the learning curves and outcome of LDP between 'pioneers' and early adopters in terms of feasibility and proficiency using short term outcomes over a period from 1997-2019.

ELIGIBILITY:
Inclusion Criteria:

* The collected data included the name of the surgeon so inclusion criteria for participating surgeons could be determined. Surgeons who were experienced with a minimum of 40 LDPs in total with at least 10 LDPs per year and who performed their LDPs in the same institution (i.e. no outside institutions) were included.

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Data of all consecutive patients who underwent elective LDP by 'pioneering' surgeons and early adopting surgeons in the period 1997-2019 were collected from a retrospective database of centers participating in the European Consortium on Minimally Invasive Pancreatic Surgery (E-MIPS) or International Consortium on Minimally Invasive Pancreatic Surgery (I-MIPS).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 1997-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Feasibility learning curve | 1997-2019
  Feasibility learning curves are based on operation time
Proficiency learning curve | 1997-2019
  Proficiency learning curves are based on major complications

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Ramshorst TME, Edwin B, Han HS, Nakamura M, Yoon YS, Ohtsuka T, Tholfsen T, Besselink MG, Abu Hilal M. Learning curves in laparoscopic distal pancreatectomy: a different experience for each generation. Int J Surg. 2023 Jun 1;109(6):1648-1655. doi: 10.1097/JS9.0000000000000408. PMID 37144678